CLINICAL TRIAL: NCT05242991
Title: Comparison of Two Photobiomodulation Protocols for the Oral Mucositis and Xerostomia Prevention in Irradiated Head and Neck Cancer Patients: a Randomized, Multicenter, Single-blind Controlled Clinical Trial
Brief Title: Effectiveness of Photobiomodulation Protocols in Radiation-induced Oral Side Effects in H&N Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: AC Camargo Cancer Center (Other); Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Manoela Domingues Martins, Associate Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PBM and MO H&N
Record Dates: First submitted 2021-12-07; First posted 2022-02-16 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Mucositis; Xerostomia; Hyposalivation
Keywords: mucositis; xerostomia; photobiomodulation; head and neck cancer; taste disorders; trismus
MeSH Terms: conditions — Mucositis; Xerostomia; Head and Neck Neoplasms; Taste Disorders; Trismus | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to one of two groups for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will not know the laser protocol of each patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intraoral photobiomodulation protocol (Active Comparator): Patients will receive the PBMT from the first day of RT, 5 times a week (Monday to Friday), for 6 to 7 weeks, or until there are no more mucositis lesions, just before the RT session. Intraoral protocol will utilize a low-level laser device (MMOptics Ltda, Sao Carlos, Sao Paulo, Brazil) with wavelength 660nm, power 100 mW, spot 0.03 cm², dose 10 J/cm², and time 3 seconds. The irradiations will be punctual and in a contact form, with 1 cm between the points, perpendicular to the oral mucosa, avoiding the tumor site and will be performed: 6 points on the labial mucosa (3 in the upper and 3 in the lower), 2 points on the labial commissure (1 on the right and 1 on the left), 8 points on the jugal mucosa (4 on the right and 4 on the left), 8 points on the lateral border of the tongue (4 on the right and 4 on the left), 5 points on the ventral tongue (2 on the right, 2 on the left side and 1 point on the apex), 4 points on the oral floor (2 on the right and 2 on the left side).
  Interventions: Device: Photobiomodulation therapy
- Extraoral photobiomodulation protocol (Active Comparator): Patients will receive the PBMT from the first day of RT, 5 times a week (Monday to Friday), for 6 to 7 weeks, or until there are no more mucositis lesions, just before the RT session.
  Extraoral protocol will utilize a defocused high-level laser device (Gemini® Diode Laser - UltraDent) with wavelength 810 + 980 nm, power 1 W, spot 4.91 cm², dose 6.11 J/cm², and time 30 seconds.
  The irradiations will be punctual and in a contact form, perpendicular to the skin, avoiding the tumor site and will be performed:
  * 5 points on the face (2 on both right and left cheeks, 2 points on both right and left parotid gland region and 1 on the lip);
  * 5 points on the neck area (1 point on the sublingual gland region, 2 points on the right and left submandibular spaces and 2 points on the neck nearby lymphatic chain).
  Interventions: Device: Photobiomodulation therapy

INTERVENTIONS:
Device: Photobiomodulation therapy — Light therapy for the management of oral side effects related to radiotherapy, mainly in the decrease of oral mucositis (OM) rates and OM severity, healing of OM ulcers and pain relief.
  Other Names: Lasertherapy

SUMMARY:
Head and neck cancer (HNC) are among the most frequent malignancies in the world. The main treatment modalities for HNC are surgical excision, radiotherapy (RT), and chemotherapy (CT). Severe oral sequelae such as oral mucositis (OM), dysgeusia, opportunistic infections, trismus, and xerostomia/hyposalivation can affect HNC patients due to oncological treatment with RT and QT. Photobiomodulation therapy (PBMT) with an intraoral low-power laser has been studied as an excellent tool in the management of OM and xerostomia and thus improves the tolerability of RT in the head and neck region. The aim of this multicenter, randomized, single-blind clinical trial is to compare the effects of two photobiomodulation protocols (intraoral application low-level laser and defocused extraoral application of high-power laser) in the management of oral mucositis (OM) and xerostomia in head and neck cancer patients undergoing radiotherapy (RT). It is expected defocused extraoral high-power photobiomodulation shows results as good as intraoral photobiomodulation on the management of oral mucositis.

DETAILED DESCRIPTION:
Radiotherapy (RT) and chemotherapy-induced oral side effects, as oral mucositis, and xerostomia are extremely challenging for professionals in the supportive care for head and neck squamous cell carcinoma (HNSCC) patients. There is a substantial evidence about the benefits of photobiomodulation in the management of these oral side effects, mainly in the decrease of oral mucositis (OM) rates and OM severity, healing of OM ulcers and pain relief by intraoral low-level lasers. However, new parameters as extraoral applications by defocused high-power lasers have been investigated to improve the OM outcomes, the patients' complaints, and the experience in the clinical assistance by professionals. Thus, 132 H&N cancer patients will be, globally and simultaneously, randomized according to clinical stage of head and neck cancer, type of treatment (isolated RT or RT and QT), type of RT (RTC3D or IMRT) and center involved (A.C. Camargo Cancer Center or State of São Paulo Cancer Institute or Porto Alegre Clinics Hospital). The randomized patients can be allocated into two groups: Group I: intraoral photobiomodulation with low level laser therapy (660nm, 100 mW, 10 J/cm2, 3 s/point) and Group II: extraoral photobiomodulation with high level laser therapy (810 + 980 nm, 1000 mW, 6.11 J/cm2, 30 s/point). PBMT will be performed daily, 5 times per week during the radiotherapy or until wound healing of OM lesions by a trained professional. Oral mucositis, pain, xerostomia, dysphagia, dysgeusia, oral functions, labial hydration and radiodermatitis will be evaluated daily. Salivary flow and trismus will be assessed weekly, and two questionaries (OHIP-14 and Vanderbilt) will be assessed on the first day of RT, on the middle of RT regimen, on the final of RT regimen and three months later RT sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of cancer in the oral cavity and oropharynx any clinical stage based on TNM staging of head and neck cancer;
* Patients who received oral care prior to oncological treatment;
* Patients who will receive conformational radiotherapy (RT-C3D) or Intensity-modulated radiotherapy (IMRT) from 50 Gy to 70 Gy (primary radiation field) in daily doses of 1.8-2, 12 Gy divided five times per week (from Monday to Friday), totalizing 6 to 7 weeks of treatment. They may receive exclusive RT or with chemotherapy concomitant with cisplatin (100 mg/m2 every 21 days or 50 mg/m2 per week);
* Patients feeding orally or by parenteral nutrition;
* Patients who agree to participate in the study after reading, filling, and signing the Consent Form for Participation in Clinical Research.

Exclusion Criteria:

* Patients who develop head and neck radiodermatitis and for this reason interrupt the survey;
* Patients who do not appear in four or more PBMT or RT sessions.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Oral mucositis | 18 months
  The measurement of mucositis will be performed daily from the first day of the radiotherapy sessions until healing by a blinded observer. Mucositis will be scored according to World Health Organization criteria: grade 0 (none), grade I (oral soreness, erythema), grade II (oral erythema, ulcers, solid and liquid diet tolerated), grade III (oral ulcers, liquid diet only), and grade IV (oral alimentation impossible).
Oral mucositis | 18 months
  The measurement of mucositis will be performed daily from the first day of the radiotherapy sessions until healing by a blinded observer. Mucositis will be scored according to the National Cancer Institute (NCI) scale (NCI - Common Terminology Criteria for Adverse Events) will be performed: grade I mucosal erythema), grade II (patchy ulcerations with pseudomembranes), grade III (confluent ulcerations or pseudomembranes, bleeding with minor trauma), and grade IV (tissue necrosis, significant spontaneous bleeding).
Ulcerated oral mucositis | 18 months
  Oral mucosal sites affected by ulcerated oral mucositis will be recorded.
Xerostomia | 18 months
  A subjective evaluation will be performed daily by a classification proposed by Eisbrush et al., 2003: grade 0 (none), grade I (), grade II (oral erythema, ulcers, solid and liquid diet tolerated), grade III (oral ulcers, liquid diet only), and grade IV (oral alimentation impossible).
Hyposalivation | 18 months
  An objective evaluation will be performed weekly by measurement and weighing of non-stimulated and stimulated salivary flow (ml/min) as proposed by Eisbrush et al., 2003.

CONTACTS AND LOCATIONS:
Overall Officials: Fábio A Alves, PhD, Principal Investigator — A.C. Camargo Cancer Center; Ana Carolina P Ribeiro e Silva, PhD, Principal Investigator — Instituto de Cancer do Estado de São Paulo; Manoela D Martins, PhD, Study Chair — Federal University of Rio Grande do Sul
Locations (1):
- Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Klein IP, Pinto MBR, So BB, de Farias Gabriel A, Mendonca NF, da Cruz Santos LB, Farias KM, Mores AL, Martins MAT, Silva ACPRE, Brandao TB, Santos-Silva AR, Alves FA, Martins MD. Intraoral vs. extraoral photobiomodulation therapy for oral mucositis in head and neck cancer patients: a multicenter, randomized, single-blind clinical trial. Support Care Cancer. 2025 Sep 10;33(10):842. doi: 10.1007/s00520-025-09877-w. PMID 40928526